CLINICAL TRIAL: NCT03501225
Title: Influence of Use of Ozonated Water in the Lower Third Molar Surgery Impacted on Pain, Swelling, Trismus, and Quality of Life.Triple Blind Randomized Clinical Trial Split Mouth
Brief Title: Effects of Ozonated Water on Pain, Swelling, Trismus and Quality of Life in Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Principal Investigator, José Cristiano Ramos Glória, Clinical professor, Federal University of the Valleys of Jequitinhonha and Mucuri
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 23032018
Record Dates: First submitted 2018-03-28; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-01

CONDITIONS: Ozone; Third Molar; Clinical Trial
MeSH Terms: interventions — Ozone; Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozone (Experimental): tooth extraction under irrigation with ozonated water
  Interventions: Procedure: ozone
- water (Experimental): tooth extraction under irrigation with ozonated water or doubly distilled water
  Interventions: Procedure: water

INTERVENTIONS:
Procedure: ozone — After local anesthesia, it was performed sulcular incision with scalpel blade number 15 and removal of soft tissues. Osteotomy was performed at low rotation and odontosecion at high speed, under constant irrigation with ozonated water. Tooth removal, careful curettage, bone regularization and surgical shop cleaning were then performed under abundant irrigation with ozonated water according to randomization. The suture was then performed.
  Arms: ozone
Procedure: water — After local anesthesia, it was performed sulcular incision with scalpel blade number 15 and removal of soft tissues. Osteotomy was performed at low rotation and odontosecion at high speed, under constant irrigation with redistilled water. Tooth removal, careful curettage, bone regularization and surgical shop cleaning were then performed under abundant irrigation with redistilled water according to randomization. The suture was then performed.
  Arms: water

SUMMARY:
The aim of this study was to evaluate the effect of ozonated water on pain, edema and trismus after third molar removal. Patients were submitted to extraction of lower third molar under irrigation with ozonated water or doubly distilled water. Data were collected at baseline, 24 hours, 48 hours, 72 hours and 7 days after intervention.

DETAILED DESCRIPTION:
The intensity of pain, the degree of edema and trismus are generally subjective and difficult to show a variation between patients. To detect this difference, we chose a split-mouth study design - one side will be assigned irrigation with ozonated water (Study Group) and the contralateral side will be assigned irrigation with double-distilled water (control group) in which each patient will be self-controled. The control side and the study side were assigned to the same patient to exclude bias from individual variations. Bias in the sample selection and evaluation of the parameters will be decreased by randomization and blinding, respectively.

Recently Resolution Conselho Federal de Odontologia (CFO) 166/2015 recognized the practice of ozone therapy by the dental surgeon. It is necessary to search for more robust and consistent results so that a careful analysis may or may not justify the routine use of ozone as a treatment modality in dentistry.

There have been no reports in literature of studies that evaluated the effects of ozonation (ozonated water), pain control, edema, trismus and quality of life, with blinding of patients, operators and evaluators, after extraction of mandibular third impacted molars. Therefore, this trial is justified in the search for new alternatives with fewer side effects in the control of postoperative complications and in the realization of a triple blind randomized clinical trial on the application of ozone in dentistry.

The main objective to evaluate the effect of the use of ozonated water on irrigation performed in bilaterally impacted and asymptomatic inferior third molars.

The secondary objectives to evaluate the quality of life in patients submitted to bilaterally impacted and asymptomatic inferior third molars and compare postoperative pain, trismus and edema in the group using ozonated water with the control side.

METHODOLOGY Study Design

A triple blind randomized controlled trial was conducted.

Location of study

Clinic of Surgery and Periodontics of the Universidade Federal dos Vales do Jequitinhonha e Mucuri (UFVJM) / Diamantina /Minas Gerais (MG)

Ethical Principles

According to resolution CNS / 12, the research project was submitted and approved by the Comitê de Ética em Pesquisa (CEP) / UFVJM (opinion nº: 2.174.074) and the study was developed according to the protocols of CONSORT.

In accordance with resolution 466 Conselho Nacional de Saúde (CNS), a presentation / explanation letter was sent to all participants, describing the main points involved in the research. Participants who agreed to the terms of the study and signed the informed consent form (TCLE-ANNEX I) were included. All participants were guaranteed surgery for extraction of lower third molars. We used the split-mouth study model (in which the patient is self-controlled), in order to exclude bias from individual variations. On one side ozonated water (as irrigating solution) was applied and on the other side, after a period of 4 weeks, double distilled water (as irrigating solution).

Sample Lectures were held about the Research Project at Tiradentes High School and Ayna Torres High School. The interested parties provided the necessary data and were later called to UFVJM for a clinical and radiographic examination.

Sample size

Sample calculation size for mean comparison (Lwanga & Lemeshow, 1991), considered the standard deviation of pain 3,32 mm (kazancioglu et al.) And the difference to be detected between groups stipulated in 3 mm, 95% significance and test power 80%, determining 19 patients. It was defined that 21 patients would be treated to avoid possible losses.

Randomization and concealment of the allocation

All extractions were pre-scheduled from January to February 2018. After establishing the inclusion and exclusion criteria, we selected 21 patients who were scheduled according to their availability for the day and time pre-established (3 surgeries per day, Monday and Tuesday in the morning: 7.30, 8.30 and 9.30). When the agenda was completed, each patient was numbered (from 1 to 21).

An independent team, (JNS) was responsible for randomization, and concealment of allocation.

The definition of which irrigating solution (double-distilled water or ozonated water) would be Protocol I or Protocol II

* the words: Protocol I and Protocol II were placed in an opaque envelope
* the words: Double-distilled Water and Ozonized Water were placed in another opaque envelope.

When making the draw it was defined that Protocol 1 would be OZONIZED WATER and obviously Protocol 2 was with DOUBLE-DISTILLED WATER.

Note: the result of the draw was revealed after the conclusion of the statistic.

For the definition of the intervention to be Protocol I or Protocol II:

* the words: Protocol I and Protocol II were placed in an opaque envelope
* the odd numbers of a dice and the even numbers of a dice were placed in another opaque envelope.

When making the draw it was defined that Protocol 1 would be any odd numbers of the dice and obviously Protocol 2 was any even numbers of the dice.

For the definition of the intervention be on the right or left side:

* the words: right side and left side were placed in an opaque envelope
* the odd numbers of a dice and the even numbers of a dice were placed in another opaque envelope.

When making the draw it was defined that the right side would be any odd numbers of the dice and obviously the left side got any even numbers of the dice.

Thus, the data was released twice for each patient. The first release corresponding to the protocol and the second release corresponding to the side to be operated. Each patient received two envelopes. For the first surgery (sequence of patients established by the schedule of surgeries), the protocol was raffled and soon after the side to be operated on was also raffled; the result was placed inside the envelope (opaque) that was duly identified with the patient's number, date, day and time (from surgery). The opposite result of the first draw was placed on the second envelope. This procedure was performed in the same way for the other 20 patients. Treatment allocation was kept secret (sealed / opaque envelopes), stored sequentially in a closet and opened only 5 minutes before each surgery in the preparation environment of the irrigating solution (Double-distilled Water and Ozonized Water).

Masking of:

* Patient: was facilitated by the fact that the procedure was performed in the mouth so the surgical tray was out of sight and the patient was wearing the peck cloth.
* Operator I (JCRG) and Assistant I (APSJ): They were "blinded" to treatment protocols (I or II). When it was time to use the irrigating solution (the JNS helper), it was taken to the surgical environment (protocol I or protocol II) in a stainless steel tank and it is poured into another stainless steel tank in the surgical tray.
* Assistant II (LDAS): performed all the measurements and applied the questionnaires, without knowing the protocols (I or II).
* Statistical (DWDO): Completed the database with all measurements and questionnaires without knowing the protocols (I or II).

Variables:

dependent variables: ozone therapy (ozonated water)

Independent variables:

A 10-sheet block containing a sequence of medications related to pain, edema and trismus was prepared for each patient. Each sheet contains the following published data: patient name, age, gender, protocol, operational side and intervention timeline, time, day of the week and data. The series was completed by Assistant II (LDAS), and there were spaces related to evaluation of edema and evaluation of buccal opening in the whole block (baseline, 24, 48, 72 hours and 7 days postoperatively) and space for evaluation of operative pain at 24, 48, 72 hours post-operatively. The measurements were individually formed, detached and placed inside one envelope so that there was influence on the result of the other.

Postoperative pain:

In order to evaluate the incidence and intensity of postoperative pain, a token was used with a visual analogue scale consisting of a horizontal line of 10 cm, with no demarcations presenting in the left extremity no pain (0), and right extremity the maximum of pain(10) (ANNEX III). The patients were instructed to mark with a vertical trace the point of the scale that best defines their degree of pain sensitivity after the surgical procedures (24, 48 and 72 hours). This marking was measured with a digital caliper (Mitutoyo® / taking into account two decimal places) by the statistician when the data was released.

Presence of edema (postoperative):

The level of facial swelling (edema) was determined by measuring with measuring tape according to the method described by angulation [27] (Photo 1). Three measures (1. measurement of the corner of the eye to the angle of the mandible, 2. measurement of the tragus at the corner of the mouth and 3. measurement of the tragus to the pogonion) were performed between the 5 reference points: tragus, pogonion lateral corner of eyes, jaw angle, outer corner of mouth. The measurements were obtained preoperatively (baseline) and in the postoperative period of 24, 48 and 72 hours and 7 days. The sum of the preoperative measurements will be the standard of normality for each side. After verification of the measurements in the postoperative period, the difference in the measurements before and after the surgical procedure was observed, determining the level of edema (APPENDIX IV).

Presence of trismus:

The maximum buccal opening will be used to assess the presence of trismus. The maximum interincisive distance was measured by the assistant II (LDAS), through a digital caliper (Mitutoyo® / taking into account two decimal places) and transcribed in millimeters for data recording. The measurement was made considering the distance between the incisal face of the right upper central incisor and the right lower central incisor after the maximum possible opening of the mouth, in the preoperative (baseline) and in the postoperative period of 24, 48 and 72 hours and 7 days. The amount of reduction of the buccal opening was measured, compared to the baseline. Thus, we calculated the relative mean between patients (Delta)

Quality of life:

After surgery, patients received the first questionnaire (Table 1) and were instructed to take it home and fill it out through the course of the week. Seven days after the surgery, the sutures were removed and the questionnaire filled with information on postoperative quality of life was collected. At that time, another questionnaire (Table 2) was completed by the patient at the clinic, after sutures were removed.

Surgery time:

The duration of the surgery was calculated through the use of a stopwatch, from the moment the incision was made until the suture. (JCRG)

Patient-related variables:

Gender, age.

Treatments

Pharmacological:

Sodium Dipyrone 500 mg and Nimesulide 100 mg

* Redistilled water (closed system of 250 ml / sterile and pyrogenic): Sanobiol laboratory.
* ozonated water (8.0 μg / ml): obtained by ozone generator philozon / medplusv, Brazil - recognized by Anvisa, coupled to the glass column with catalytic converter and microbubble diffuser in stainless steel tube. According to Nogales CG et al (2014), water (double-distilled) does not absorb all the concentration offered to it. This ratio is between 20 and 25% absorption. In this sense, the ozone generator was regulated at 40mcg (40 μg/ml) for 5 (five minutes) of bubbling in 250 ml of doubly distilled water to obtain 8.0 μg / mL ozone / water concentration. An ozonated water was prepared for each surgery and used immediately.

Surgical procedure Antisepsis and local anesthesia

For the extraoral antisepsis we used an alcoholic solution of 10% polyvinylpyrrolidone-iodine (PVP-I). For local anesthesia, the technique of regional inferior and lingual alveolar nerve block was used, with complementation of the buccal nerve anesthesia, with the care of slow injection of the solution, after negative aspiration. For each surgery a maximum volume of up to 5.4 mL of local anesthetic solution containing 2% lidocaine and 1: 100,000 epinephrine (equivalent to 3 tubes of a local anesthetic solution) was used.

Surgical intervention The surgical procedures were performed in two sessions, with a 30-day interval for each side of the hemimandible and the choice of the side to be operated in the first session was random. Mandibular third molar surgeries were performed by a professional with experience in this type of intervention and he was blind as to the type of treatment that the patient underwent.

The surgical technique used for all cases can be described as follows: after incision of Avellanal (1946) with a scalpel blade number 15 and separation of soft tissues for surgical site exposure, a low rotation osteotomy (30,000 rpm) was performed with drill bit 8 mounted on straight handpiece and high-speed drill 350,000 rpm with 702 C KG Sorensen carbide drills mounted on a Dabi Atlante® high-speed handpiece at 350,000 rpm under constant irrigation with (double-distilled water or ozonated water according to randomization) .

Then, the tooth extraction was performed with the aid of straight elevators of the Seldin type, careful curettage, bone regularization and cleaning of the surgical area by means of abundant irrigation with (double-distilled water or ozonated water according to the randomization). The suture was performed with silk thread (4.0) through isolated stitches. Hand-irrigation of double-distilled water or ozonated water (packed in small steel vats) was performed with the use of a 10cc hypodermic glass syringe (ruthe brand) attached to a 10mm (BD mark) steel needle.

The patients were re-evaluated (24.48.72 hours and 7 days for edema and trismus and 24.48.72 hours for pain intensity) after surgery, by an investigator (assistant II / LDAS) who was "blinded" about the type of intervention that the patient underwent. In addition to the removal of the suture on the 7th day, this same researcher collected and applied the quality of life questionnaires.

Biosafety procedures

National biosafety standards and recommendations were followed for both infection control and waste disposal. Operator I was responsible for maintaining adequate infection control during clinical examination and surgery procedures. The assistant II was responsible for the same control in the postoperative evaluations. The researchers conducted the examinations and evaluations wearing white clothing, hat, mask, white apron and disposable latex gloves. The instruments used were sterilized by autoclave.

Data processing

The results were typed and organized into a database, using the software Statistical Package for Social Science (SPSS), version 23.0. Processing included encoding, typing and editing data. This process was performed by two people, (one typed the data and the other checked the data that was typed). Each envelope containing the data of each patient received a corresponding number in the database.

Statistical analysis of data

A descriptive analysis was performed of the absolute and relative frequencies of all the variables studied and the association tests. The data according to the different types of intervention will be analyzed through the t-student test and the Wilcoxon test. The level of significance will be p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* impacted lower third molar
* class II-B of Pell-Gregory classification
* No systemic disease

Exclusion Criteria:

* local infection
* previous periocoronaritis
* smoke
* allergy to ozone

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain at 72 hours | 24hours, 48hours, 72hours
  Post-operative pain measured by visual analogic scale (VAS). The VAS comprises a 10cm horizontal line, with no marks. When responding to a VAS, subjects specify their level of pain by indicating a position along a continuous line between two end-points. Higher values represent a worse outcome.
Change from Baseline Swelling at 7 days | baseline, 24hours, 48hours, 72hours, 7 days
  post-operative swelling measured from tragus to mouth corner
Change from Baseline trismus at 7 days | baseline, 24hours, 48hours, 72hours, 7 days
  maximum mouth opening measured as maximum distance between incisal edges of upper and lower central incisors.

SECONDARY OUTCOMES:
Change from Baseline Quality of life at 7 days | baseline, 7 days
  Oral health related quality of life measured by questions related to the quality of life. This questionnaire comprises 22 items within 6 subscales (social isolation, working isolation, eating ability, speaking ability, sleep impairment, physical appearance). The questions should be responded as yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: José Cristiano Ramos Glória, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri
Locations (1):
- Universidade Federal dos Vales do Jequitinhonha e Mucuri, Diamantina, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gloria JCR, Douglas-de-Oliveira DW, E Silva LDA, Falci SGM, Dos Santos CRR. Influence of ozonized water on pain, oedema, and trismus during impacted third molar surgery: a randomized, triple blind clinical trial. BMC Oral Health. 2020 Feb 5;20(1):41. doi: 10.1186/s12903-020-1029-5. PMID 32024498